CLINICAL TRIAL: NCT01347658
Title: DRUG INTERACTIONS BETWEEN ECHINACEA PURPUREA AND ETRAVIRINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECHI-ETRA
Record Dates: First submitted 2011-03-22; First posted 2011-05-04 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2011-09

CONDITIONS: HIV
Keywords: etravirine; Echinacea purpurea; interaction
MeSH Terms: interventions — Echinacea extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etravirine + echinacea (Experimental): etravirine + root of Echinacea purpurea
  Interventions: Dietary Supplement: Echinacea purpurea

INTERVENTIONS:
Dietary Supplement: Echinacea purpurea — Patients will take Echinacea purpurea (500 mg every 8 hours) during 14 days.

SUMMARY:
The purpose of this clinical trial is to characterize drug interactions between one medicinal herb: Echinacea purpurea and the protease inhibitor etravirine.

DETAILED DESCRIPTION:
Because of its CYP3A4 inducer activity in the liver but its inhibitor effect at the intestinal site, concomitant administration of Equinacea purpurea (a medicinal herb frequently used by HIV-infected patients) and etravirine (an HIV reverse transcriptase inhibitor) might result in clinically relevant pharmacokinetic drug interactions.

15 HIV-infected patients on stable antiretroviral therapy including etravirine at the dosage of 200 mg twice daily during at least 4 weeks will be enrolled. After their inclusion in the study, patients will receive Echinacea purpurea root (500 mg every 8 hours) in addition to their antiretroviral treatment, from day 1 until two weeks later (day 14). On days 0 and 14, blood samples will be drawn immediately before and 1, 2, 4, 6, 8, 10 and 12 hours after the administration of an etravirine dose, and etravirine concentrations in plasma will be determined by high performance liquid chromatography using a validated method.

ELIGIBILITY:
Inclusion criteria:

1. Patients infected with HIV-1 (at least one documented positive Western-Blot).
2. Age 18 years or more.
3. Patients receiving antiretroviral therapy including etravirine at the approved dose of 200 mg twice daily for at least 4 weeks
4. HIV viral load in plasma <50 copies / mL
5. Absence of acute infections and / or tumors in the three months prior to inclusion.
6. Subject able to follow the treatment period, without suspicion of poor adherence in previous antiretroviral treatments.
7. Voluntary written informed consent.

Exclusion criteria:

1. Any clinical or historical observation that could interfere with the pharmacokinetics of medications, such as gastrointestinal illness or surgery (except for herniotomy and appendectomy), changes in the composition of plasma proteins, some indication of hepatic or renal dysfunction.
2. Antiretroviral regimen including drugs ritonavir or atazanavir (CYP3A4 inhibitors)
3. Concomitant treatment with drugs inductors of CYP3A4 (rifampicin, fenitoin, carbamazepin, ...)
4. Active alcohol consumption (> 50 g / day) or illicit drugs (except cannabis).
5. Pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
plasma concentration of etravirine. | Change from baseline to day 14
  plasma concentration of etravirine.

SECONDARY OUTCOMES:
Clearance (CL/F) | Change from baseline to day 14
Volume of distribution (V/F) | Change from baseline to day 14
Elimination half-life (t1/2) | Change from baseline to day 14
Area under the plasma concentration-time curve during the dosing interval (AUC0-24) | Change from baseline to day 14
Number of patients with adverse events | From baseline to day 28
HIV Viral load in plasma | Day 14
Number of patients with laboratory alterations | From baseline to day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain